CLINICAL TRIAL: NCT00504725
Title: Ketamine In Thoracic Surgery (KITS) Trial
Acronym: KITS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00000895
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Results first posted 2012-11-16 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2012-11

CONDITIONS: Lung Cancer
Keywords: Lobectomy; VATS
MeSH Terms: conditions — Lung Neoplasms | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Experimental): Single bolus 0.5mg/kg ketamine IV after induction of anesthesia
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): 0.9 % saline bolus of equivalent volume
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: Ketamine — Interventional
  Arms: Ketamine
Drug: 0.9% saline — placebo
  Arms: Placebo

SUMMARY:
The primary aim of the study is to demonstrate a reduction in circulating interleukin 6 levels at 4 and 24 hours after completion of lobectomy (either VATS or open). The null hypothesis (H0) is thus that there is no difference in circulating interleukin 6 levels when patients are given either ketamine or placebo (0.9% saline in equivalent volume). The alternative (two tailed) hypothesis (HA) if the null is disproved is that ketamine leads to significantly different levels of interleukin 6 at 4 and 24 hours after completion of surgery. We plan to randomize 40 patients to receive either ketamine or placebo, in a block of 4 randomization design stratified by whether surgery is performed by VATS or open lobectomy.

DETAILED DESCRIPTION:
This study is designed to be a phase 2 (efficacy) randomized controlled clinical trial of ketamine versus placebo in 40 patients undergoing lobectomy by VATS or open approach, at Duke University. We selected a single dose regimen of 0.5mg/kg IV ketamine given at induction of anesthesia, as this is the dose that previously has been shown to induce maximal suppression of the IL-6 response in cardiac surgery.

We plan to randomize 40 patients to receive either ketamine or placebo, in a block of 4 randomization design stratified by whether surgery is performed by VATS or open lobectomy. 40 patients (n=20 per group) will provide 90% power to detect a change in IL 6 of 20 pg/ml from a mean of 100 pg/ml at 4 hours, with two tailed alpha = 0.05. Allowing for 10-20% attrition we will enroll 50 patients to achieve this sample size. All patients presenting for lobectomy either VATS or open will be included. Patients will be screened by review of the preoperative surgical schedule posted each day and approached for consent to participate if they do not have any exclusion criteria. Patients who are randomized but do not undergo lobectomy for any reason will not be included in the analysis of the primary endpoint. Patients who are listed for VATS resection but convert to open will be included in the analysis on a per protocol basis. The randomization is stratified according to planned approach (VATS vs open), however we expect the majority of these cases to be VATS lobectomies.

Treatment will be by intravenous administration of a single dose of study drug over 5 minutes immediately after induction of anesthesia and before surgical incision.

Patients will be randomized (by sealed envelope) in blocks of 4 to receive ketamine or placebo. The randomization will be stratified according to whether the planned surgery is via VATS or open (thoracotomy) approach. The study drug will be prepared by the investigational pharmacy and provided to the attending anesthesiologist of record for the case. It will contain 0.5 mg/kg ketamine for injection by IV bolus over 5 minutes, or as an equivalent volume of 0.9% saline. It will be the responsibility of the principal investigator to ensure that study drug is administered in a timely fashion, usually by delegation to the attending anesthesiologist of record for the case. The anesthetic procedure will be standardized in that each patient will receive a total intravenous anesthetic using propofol and an intravenous opioid infusion. This anesthetic will be supplemented by an epidural and intravenous opioid boluses as needed to control pain.

Visits by the research team will be performed as follows:

1. Visit 1 will occur at enrollment, when baseline information (see CRF visit 1) will be collected and study consent forms signed.
2. Visit 2 will occur at induction of anesthesia when study drug will be administered and a baseline blood sample of 10ml collected from the patient's arterial line. The blood sample will be immediately centrifuged and the serum frozen and stored for subsequent analysis.
3. Visit 3 will occur at 4 hours after completion of surgery when 10 ml blood will be collected and CRF visit 3 form will be completed (VAS score and emergence delirium).
4. Visit 4 will occur at 24 hours after completion of surgery when 10 ml blood will be collected and CRF visit 4 form will be completed (VAS score).
5. The final visit will occur just prior to hospital discharge when CRF visit 5 form will be completed (secondary endpoints). Additionally, if the principal investigator is informed by either study staff or the clinical team of an adverse event or other complication, then the patient will be visited within 24 hours for confirmation of the event and ascertainment of whether the event is related to study drug or not. An SAE form will be completed and sent to the IRB in line with institutional policy.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting for lobectomy either VATS or open.

Exclusion Criteria:

* Patients with myocardial infarction in the previous six months,
* Patients with a history of psychotic disorder,
* Patients with a history of chronic pain syndrome,
* Patients with documented previous allergy to ketamine.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andy Shaw, M. D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Roytblat L, Talmor D, Rachinsky M, Greemberg L, Pekar A, Appelbaum A, Gurman GM, Shapira Y, Duvdenani A. Ketamine attenuates the interleukin-6 response after cardiopulmonary bypass. Anesth Analg. 1998 Aug;87(2):266-71. doi: 10.1097/00000539-199808000-00006. PMID 9706914
- [Background] Bartoc C, Frumento RJ, Jalbout M, Bennett-Guerrero E, Du E, Nishanian E. A randomized, double-blind, placebo-controlled study assessing the anti-inflammatory effects of ketamine in cardiac surgical patients. J Cardiothorac Vasc Anesth. 2006 Apr;20(2):217-22. doi: 10.1053/j.jvca.2005.12.005. Epub 2006 Mar 9. PMID 16616662 (Retraction: PMID 25319992 J Cardiothorac Vasc Anesth. 2014 Oct;28(5):1435)
- [Background] Tashima T, Yamashita J, Nakano S, Joutsuka T, Hayashi N, Saishoji T, Ogawa M. Comparison of video-assisted minithoracotomy and standard open thoracotomy for the treatment of non-small cell lung cancer. Minim Invasive Ther Allied Technol. 2005;14(3):203-8. doi: 10.1080/13645700510034001. PMID 16754164
- [Background] Craig SR, Leaver HA, Yap PL, Pugh GC, Walker WS. Acute phase responses following minimal access and conventional thoracic surgery. Eur J Cardiothorac Surg. 2001 Sep;20(3):455-63. doi: 10.1016/s1010-7940(01)00841-7. PMID 11509263
- [Background] Yim AP, Wan S, Lee TW, Arifi AA. VATS lobectomy reduces cytokine responses compared with conventional surgery. Ann Thorac Surg. 2000 Jul;70(1):243-7. doi: 10.1016/s0003-4975(00)01258-3. PMID 10921716

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine | Placebo
Started | 21 | 20
Completed | 20 (Prior to unblinding, one subject was discontinued due to elevated CRP levels at baseline.) | 20
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Placebo | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: Years]
  AGE | 61 (12) | 66 (10) | 63 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 11 | 12 | 23
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Interleukin Levels at 24 Hours
Time Frame: 24 Hours
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 20 | 20
pg/ml
  Interleukin-6 (IL-6) | 245 (287) | 269 (210)
  Interleukin-8 (IL-8) | 11.3 (12.6) | 14.8 (10.8)
  Interleukin-10 (IL-10) | 3.0 (4.7) | 4.9 (5.8)
Statistical Analysis 1: Comparison: Ketamine vs Placebo; IL-6; Test type: Superiority or Other; p = 0.39, ANOVA — We will use two way ANOVA (looking for effects due to drug and time) with a p value of 0.05 indicative of statistical significance
Statistical Analysis 2: Comparison: Ketamine vs Placebo; IL-8; Test type: Superiority or Other; p = 0.18, ANOVA
Statistical Analysis 3: Comparison: Ketamine vs Placebo; IL-10; Test type: Superiority or Other; p = 0.14, ANOVA

2. Secondary Outcome: C-reactive Protein (CRP) Serum Levels
Description: The CRP levels were measured 24 hours postoperatively.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 20 | 20
pg/ml | 8.8 (4.5) | 9.3 (5.6)
Statistical Analysis 1: Comparison: Ketamine vs Placebo; Test type: Superiority or Other; p = 0.37, ANOVA

3. Secondary Outcome: Verbal Pain Scores
Description: Pain scores rated by the subject on a scale of 0 low - 10 high
Time Frame: baseline, 4 hours, 24 hours and at discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 0.30 (0.73) | 0.35 (1.35)
  4 Hours | 3.8 (2.1) | 3.1 (2.8)
  24 Hours | 2.6 (2.2) | 2.8 (2.1)
  Discharge | 1.8 (2.5) | 1.1 (1.8)
Statistical Analysis 1: Comparison: Ketamine vs Placebo; Test type: Superiority or Other; p = 0.44, Fisher Exact — Baseline Pain Level Score
Statistical Analysis 2: Comparison: Ketamine vs Placebo; Test type: Superiority or Other; p = 0.20, Fisher Exact — 4 Hour Pain Level Score
Statistical Analysis 3: Comparison: Ketamine vs Placebo; Test type: Superiority or Other; p = 0.37, Fisher Exact — 24 Hour Pain Level Score
Statistical Analysis 4: Comparison: Ketamine vs Placebo; Test type: Superiority or Other; p = 0.15, Fisher Exact — Pain Level Score at Discharge

ADVERSE EVENTS:
Arm/Group | Ketamine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 6/20 | 5/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=20) | Placebo (N=20)
AF (Cardiac disorders) | 3 (3) | 3 (3)
CHEST TUBE PLACEMENT (Surgical and medical procedures) | 1 (1) | 1 (1)
SMALL BOWEL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
RESPIRATORY INSUFFICIENCY (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No